CLINICAL TRIAL: NCT06632509
Title: BD SiteRite(TM) 9 Ultrasound System - Clinical Study
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: MDS-23SITERITE001
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: BD SiteRite 9 for VAD Insertion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- USGVAD: Patient who is a candidate for an ultrasound-guided vascular access device (USGVAD) placement procedure using SiteRite 9 System as assessed per their clinician(s)
  Interventions: Device: BD SiteRite(TM) 9

INTERVENTIONS:
Device: BD SiteRite(TM) 9 — Ultrasound-guided vascular access device placement procedure using the BD SiteRite(TM) 9.

SUMMARY:
This post-market study is being conducted to generate safety and performance data on the SiteRite 9 System. The data will be utilized to support regional registrations (for example, EU MDR), and document any unforeseen residual risks.

DETAILED DESCRIPTION:
This is an observational post-market, human subject study to evaluate the safety and performance of the SiteRite 9 System. Subjects will be recruited for participation based on need for Vascular Access Device (VAD) placement in a hospital setting.

Enrolled subjects will go through ultrasound-guided Vascular Access Device (USGVAD) placement as part of their clinical care. USGVAD is defined as a procedure in which an ultrasound machine is used to assist a qualified health care provider with IV cannulation from skin puncture through venipuncture via direct visualization on the ultrasound machine in real time.

ELIGIBILITY:
Inclusion Criteria

* Age 1 years, or older
* A patient who is a candidate for an ultrasound-guided VAD placement procedure using SiteRite 9 System as assessed per their clinician(s)
* Able and willing to provide informed consent or legal authorized representative (LAR) authorized to give consent on behalf of the subject

Exclusion Criteria:

* Any patient in whom ultrasound procedure might interfere with medical care or create undue hardship
* Known, or suspected, allergy to materials contained in the SiteRite 9 System or accessories that may come in contact with the patient
* Localized skin, tissue, or other clinical factors that would prevent completion of the ultrasound procedure
* Previous medical history that would prevent completion of the ultrasound procedure

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects are defined as patients who need to receive insertion of a vascular access devices (VAD) as part of their medical treatment.
Sampling Method: Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Primary Performance: To provide visualization of the target vessel in which to insert the chosen vascular access device. | During the procedure
  The BD SiteRiteTM 9 Ultrasound System is able to visualize the target vasculature (>=70% with a 95% confidence interval)
Primary Performance: To have successful vascular access either by cannulation or blood return. | During the procedure
  Successful access with the vascular access device, either by cannulation or blood return (>=70% with a 95% confidence interval)
Primary Safety: To determine the incidence of device related adverse events, experienced by patient or user, when using the BD SiteRiteTM 9 Ultrasound System. | During the procedure and 15 minutes after the procedure
  Rate of device related adverse events (<2%).

CONTACTS AND LOCATIONS:
Locations (1):
- Brookdale University Hospital & Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No